CLINICAL TRIAL: NCT01574911
Title: Development and Validation of a Limb Volumetry Technique Applicable in Daily Clinical Practice Using Self Positioning 3D Laser Scanning:Reproductibility and Comparison to the Reference Method
Brief Title: Validation of a New Method of Limb Volumetry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF8834
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Edema; Chronic Venous Insufficiency; Lymphedema
Keywords: volumetry 3D; Displacement of water; lymphoedema; Venous chronic insufficiency
MeSH Terms: conditions — Edema; Lymphedema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Validation study an innovative non-invasive diagnostic technique. Biomedical research conducted with the help of Montpellier University Hospital Clinical Investigation Center (CIC) for the recruitment of healthy controls, and vascular Medicine clinics for the recruitment of patients with chronic venous insufficiency or lymphedema
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- healthy adults: The objective of this project is the validation of real time reconstruction and calculation of limb volume using a 3 D laser scanner In each subject limb volume will be measured once by water - displacement and twice by 3D laser scanning
- Adults Chronic venous insufficiency: The objective of this project is the validation of real time reconstruction and calculation of limb volume using a 3 D laser scanner In each subject limb volume will be measured once by water - displacement and twice by 3D laser scanning
- patients primary lymphedema: The objective of this project is the validation of real time reconstruction and calculation of limb volume using a 3 D laser scanner In each subject limb volume will be measured once by water - displacement and twice by 3D

SUMMARY:
Volumetry is essential for the diagnosis and follow-up of patients with limb edema. The objective of this project is the validation of real-time reconstruction and calculation of limb volume using a 3D laser scanner.

Water - displacement volumetry (water-filled boot) is the reference method with known accuracy and reproducibility, but is not commonly used in clinical practice because it is cumbersome, difficult, and time-consuming. The most commonly used method remains segmental limb perimetry with a tape measure, followed by volume calculation using the truncated cones formula, thus excluding de facts extremities (hands and feet) which can neither be likened to cones nor easily measured.

Quantification limb volume and volume changes is essential for the diagnosis and follow-up of patients with chronic venous insufficiency or lymphedema, two very common pathological conditions. It is mandatory for the evaluation of therapeutic approaches.

The present study will use an innovative technology of volume acquisition by freehand laser scanning with a hand-held camera with Quantification limb volume and volume changes is essential for the diagnosis and follow-up of patients with chronic venous insufficiency or lymphedema, two very common pathological conditions. It is mandatory for the evaluation of therapeutic approaches.

The present study will use an innovative technology of volume acquisition by freehand laser scanning with a hand-held camera with real-time 3D reconstruction.

Its advantages are non-contact, accurate and detailed quantification of edema, including extremities, allowing to assess the magnitude and topography of physiological, pathological, or treatment - induced volume changes. This approach will ultimately provide data that will used for designing personalized limb compression ortheses.

DETAILED DESCRIPTION:
In each subject and patient, limb volume will be measured once by water - displacement (WD) and twice by 3D laser scanning (3D), by 2 independent operators, in random order. In a subgroup of patients, measurements will be repeated in the morning and evening, twice a year (during winter and during summer) to estimate the nycthemeral and seasonal effects.

Measurements will be performed in healthy subjects and in patients with chronic venous insufficiency or lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Either healthy adult or - Adult and chronic venous insufficiency C1s, C3, or C5 (CEAP classification) or - Primary lymphedema (between 10-90 years old)

Exclusion Criteria:

* No consent form

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment of healthy controls and vascular Medicine clinics for the recruitment of patients with chronic venous insufficiency or lymphedema
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Difference between limb volume measured | 36 months
  Difference between limb volume measured during the same session by water displacement and by 3D laser scanner

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Montpellier, Montpellier, Herault, France